CLINICAL TRIAL: NCT00411398
Title: A 10 Week Open-Label Pilot Study to Evaluate the Effectiveness and Safety of Memantine(Namenda) as Augmentation Therapy in Patients With Generalized Anxiety Disorder (GAD) or Social Anxiety Disorder (SAD), Who Are Only Partial Responders to Selective Serotonin-Norepinephrine Reuptake Inhibitors (SNRI's) or Selective Serotonin Reuptake Inhibitors (SSRI's).
Brief Title: A 10 Week Open-Label Pilot Study to Evaluate the Effectiveness and Safety of Memantine(Namenda) as Augmentation Therapy in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Thomas L. Schwartz, M.D., Assoc Professor, State University of New York - Upstate Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAM-MD-46; IRB # 5343
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: General Anxiety Disorder, Social Anxiety Disorder
Keywords: Anxiety, SNRI, SSRI,GAD,SAD
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Anxiety Disorders | interventions — Memantine

ARMS (1):
- Memantine 5-20mg/d flexible dose (Experimental): Memantine tablets 5-20mg/d flexible dose
  Interventions: Drug: Namenda/Memantine

INTERVENTIONS:
Drug: Namenda/Memantine — 5mg tablets, 1-4 tabs by mouth per day

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of memantine Add-On treatment of patients who are currently taking an SNRI or SSRI and who remain anxious and symptomatic despite treatment.

Secondary objectives of this study are:

•-to evaluate if there is an improvement in disability levels following memantine dosing

-to evaluate if there is an improvement in sleep quality following memantine dosing

DETAILED DESCRIPTION:
Memantine is an FDA approved treatment which helps slow down the progression of Alzheimer's dementia.. It is felt that high glutamate levels associated with Alzheimer's dementia are toxic to neurons which ultimately die off causing the dementia process to continue. Memantine partially blocks the NMDA glutamate channels located on neurons in the brain. This way, if glutamate rises, its toxic activity is blunted and neurons tend to become less toxic and suffer less atrophy and death.

Glutamate is felt to play a role in the development of anxiety as well. Glutamate is often in balance with another neurotransmitter, GABA. This GABA-glutamate balance (when GABA is low and Glutamate is normal to high) is also felt to play a role in the development of GAD or SAD. Low GABA and high glutamate levels (similar to the state of alcohol withdrawal) are implicated in causing anxiety symptoms. Sometimes, GABA-increasing sedative drugs, such as diazepam (Valium) are used to raise GABA activity to ward of anxiety symptoms and create a better balance between the stimulatory glutamate and inhibitory GABA. Given memantine's ability to lower glutamate levels, it may be able to also lower anxiety without the need for a sedative medication. Lowering glutamate this way, may allow a patient's own GABA concentrations to be more effective in lowering GAD or SAD symptoms.

The usual treatment in initial treatment for anxiety is to use a serotonin neurotransmitter enhancing drug, such as paroxetine or escitalopram. These 'SSRI' drugs, unlike the sedatives noted above, do not have addiction potential and are safer to use. In the anxiety disorder population, only 30-70% of patients achieve full remission of anxiety symptoms when placed on SSRI monotherapy. The usual second-line choice is to treat with a serotonin-norepinephrine enhancing SNRI, such as venlafaxineXR in order to achieve remission. If resistance occurs to the SNRI, to promote full anxiety symptom relief, addition of a GABA enhancing-sedative (to raise GABA balance) to the SNRI is a reasonable polypharmacy strategy. Sedatives, like alprazolam, are addictive and considered third line agents now. The authors feel that memantine, given its ability to manipulate the GABA-glutamate balance by lowering glutamate without major side effects (weight gain, sexual problems, (ie SSRI/SNRI) nor addiction (ie sedatives) may be a reasonable add-on or augmentation strategy to better alleviate anxiety in SNRI or SSRI partial responders.

This study is designed to evaluate generally or socially anxious patients who are only partially responsive to typical SNRI or SSRI anti-anxiety medication therapy. Patients who are less than 50% anxiety-alleviated on their SNRI medication will be asked to join the study and be placed on memantine as well. This type of add-on therapy is common in outpatient psychiatric care. This is a rater-blinded, patient open-label, non-placebo prospective pilot study, where all subjects will receive memantine for 10 weeks. This study would be the first to date in this treatment-resistant patient population, as the investigators will utilize the most comprehensive set of rating scales to date in order to best categorize patient responses in regards to anxiety with this drug.

ELIGIBILITY:
Inclusion Criteria:Patients are included in the study if all of the following criteria are met:

1. Written informed consent is obtained.
2. The patient is English-speaking and18 through 64 years of age inclusive.
3. The patient meets the DSM-IV criteria for generalized anxiety disorder or social anxiety disorder as determined by the MINI and psychiatric evaluation.
4. The patient is currently taking venlafaxine XR- SNRI or a SSRI medication for ≥ 6 weeks and on a stable, adequate therapeutic dosage and remains anxiety symptomatic
5. The patient has a total score of at least 10 on the HAM-A scale
6. The patient has a score of at least 5 on the HADS anxiety subscale score at the screening and baseline visits.
7. The patient has a CGI-S showing that anxiety symptom burden is impacting negatively on subject's life
8. The patient is in good health as determined by a medical and psychiatric history, medical examination, and cannot have major medical illness that would jeopardize patient health during the study.
9. Women must be of nonchildbearing potential [i.e., postmenopausal, be surgically sterile (hysterectomy or tubal ligation)] or must meet all of the following conditions: using a reliable, medically accepted form of contraception for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; and adequate barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen). Women must be given a pregnancy test (ßHCG), unless they are at least 2 years postmenopausal or surgically sterile, and the results of the test must be negative.
10. The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

Patients are included in the study if all of the following criteria are met:

1. Written informed consent is obtained.
2. The patient is English-speaking and18 through 64 years of age inclusive.
3. The patient meets the DSM-IV criteria for generalized anxiety disorder or social anxiety disorder as determined by the MINI and psychiatric evaluation.
4. The patient is currently taking venlafaxine XR- SNRI or a SSRI medication for ≥ 6 weeks and on a stable, adequate therapeutic dosage and remains anxiety symptomatic
5. The patient has a total score of at least 10 on the HAM-A scale
6. The patient has a score of at least 5 on the HADS anxiety subscale score at the screening and baseline visits.
7. The patient has a CGI-S showing that anxiety symptom burden is impacting negatively on subject's life
8. The patient is in good health as determined by a medical and psychiatric history, medical examination, and cannot have major medical illness that would jeopardize patient health during the study.
9. Women must be of nonchildbearing potential [i.e., postmenopausal, be surgically sterile (hysterectomy or tubal ligation)] or must meet all of the following conditions: using a reliable, medically accepted form of contraception for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Reliable forms of contraception include oral, implanted, or injected contraceptives; intrauterine devices in place for at least 3 months; and adequate barrier methods in conjunction with spermicide (abstinence is considered an acceptable contraceptive regimen). Women must be given a pregnancy test (ßHCG), unless they are at least 2 years postmenopausal or surgically sterile, and the results of the test must be negative.
10. The patient must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period, and willing to return to the clinic for the follow-up evaluation as specified in this protocol.

    -

Exclusion Criteria: Patients are excluded from participating in this study if 1 or more of the following criteria are met:

1. The patient is on more than one antidepressant or anxiolytic as a standing dose. PRN use of anxiolytic or sleeping agents may be continued at discretion of the investigator
2. The patient has an active substance misuse disorder
3. The patient is a significant risk of suicide
4. The patient has recently started psychotherapy or counseling (within last 6 weeks)
5. The patient has other psychiatric Axis-I disorders as a principal diagnosis (except generalized anxiety) within 6 months of screening and baseline visits; any history of OCD, psychotic disorder, bipolar disorder, mental retardation, or clear personality disorder. Patient may have a co-morbid substance misuse, depressive or anxiety disorder if it has been in remission for at least 6 months prior to screening visit.
6. The patient has previously participated in any clinical study are has been treated with memantine or venlafaxine XR.
7. The patient has used an investigational drug within 1 month before the screening visit or is participating in a concurrent clinical trial.
8. The patient has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery).
9. The patient is unlikely to comply with the study protocol, be unreliable in providing ratings, or is unsuitable for any reason, as judged by the investigator.
10. The patient has a clinically significant deviation from normal in the physical examination.

    -

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Schwartz, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University Psychiatry Dept., Syracuse, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects were recruited easily by radio and newspaper advertisements
Groups:
- Memantine: Memantine tablets
Period: Overall Study
Arm/Group | Memantine
Started | 15
Completed | 10
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Scale
Description: Standard Clinical Depression Rating Scale. Clinician administered. Scale units are points/numbers. Possible range is 0 to 44 with the latter signifying more severe anxiety
Time Frame: 10 wk
Population: LOCF if at least one post baseline visit completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 10
units on a scale | 10.9 (2.04)

ADVERSE EVENTS:
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=15)
nausea (Gastrointestinal disorders) | 3 (3)
headache (Nervous system disorders) | 3 (3)
Fatigue (General disorders) | 2 (2)
Edema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No